CLINICAL TRIAL: NCT01783379
Title: Pharmacokinetics of Micafungin (Mycamine ®) Given Intravenously as Therapy to Patients With an Invasive Fungal Infection in the Intensive Care Unit - a Search for Co-variates
Brief Title: Pharmacokinetics of Micafungin in Patients Intensive Care Unit
Acronym: MIMIC
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCN AKF 12.05
Record Dates: First submitted 2013-01-09; First posted 2013-02-04 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Invasive Fungal Infection
Keywords: invasive fungal infection; micafungin; intensive care; pharmacokinetics
MeSH Terms: conditions — Invasive Fungal Infections | interventions — Micafungin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples for pharmacokinietic analysis will be collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICU patient on micafungin: ICU patients with an invasive fungal infection on micafungin treatment
  Interventions: Drug: micafungin

INTERVENTIONS:
Drug: micafungin — 100mg/day infusion in 1 hour
  Other Names: Mycamine

SUMMARY:
In this trial, our goal is to determine the pharmacokinetics of micafungin in a non-selected cohort of patients with suspected or proven invasive fungal infections. Patients will receive micafungin for the period necessary to achieve clinical and / or mycological cure. An attempt will be made to have 2 PK curves, one full and one limited sampling on days 3 (n=9) and 7 (n=5). Furthermore, we will be able to determine intra-individual variability. On non-PK days, trough samples will be taken to determine the time to steady state. All samples will be taken just prior to the morning dose of micafungin. All infusion rates will be according to the SPC label information. Patients are considered to be evaluable if at least the first PK curve has been completed. Two moments of PK analysis will enable us to determine whether there is an increase over time in exposure if steady state has not been reached.

DETAILED DESCRIPTION:
Whilst micafungin (Mycamine®) has much to offer, little is known about its pharmacokinetic profile in ICU patients with specific co-morbidities such as obesity, hypoalbumenia, and severe liverfunction disturbances. Also, ICU patients are known to experience changes in pharmacokinetics (PK) due to changes in hemodynamics, extracorporeal elimination techniques, interacting comedication, etc. Based on criteria outlined below, micafungin may prove to be the drug of choice in this cohort of patients. Therefore it seems prudent to conduct a trial in a cohort of patients who receive micafungin but with co-variates that may be of influence to the pharmacokinetic profile. To build a valid pharmacokinetic model, all patients on micafungin will be included in the analysis and used for model building. Co-variates that will be explored are at least: obesitas, liverfunction, albumin, creatinin-clearance. Simulations will be performed to determine if adequate exposure is reached under different patho-physiological conditions.

In conclusion: this trial is on determining the PK of micafungin in a non-selected cohort of patients with suspected or proven invasive fungal infections. Most important covariates will be modelled using advanced mathematical techniques. Micafungin may prove to be beneficial over the other two echinocandins in terms of limited factors that impact PK. This has to be proven in a prospective trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is admitted to an ICU
2. Subject is at least 18 years of age on the day of the first dosing
3. If subject is female: neither pregnant nor able to become pregnant and is not nursing an infant
4. Subject has been treated with micafungin for a maximum of two days before enrolment in this trial
5. Is managed with a central venous catheter or an arterial catheter

Exclusion Criteria:

1. Is known to be hypersensitive to echinocandin antifungal agents
2. Documented history of sensitivity to excipients similar to those found in the micafungin preparation
3. Known of positive HIV test or positive hepatitis B or C test in history
4. History of or current abuse of drugs, alcohol or solvents
5. Has previously participated in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients receiving micafungin for the treatment or suspicion of an invasive fungal infection will be included. At least 20 patients will be included to obtain 16 evaluable patients. If recruitment of 20 patients is achieved within one year, more patients can be included. A formal sample size cannot be performed for several reasons but the sample size is rather based on the general assumption that 16 patients are sufficient to have a descriptive PK approach.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
micafunigin AUC | Day 3 and Day 7
  AUC0-tau [mg*g/L] of micafungin given to ICU patients. Other pharmacokinetic parameters will be assessed as well.

SECONDARY OUTCOMES:
covariates | 17 days
  co-variates of influence on the pharmacokinetics of micafungin. Specific co-variates are of high interest to the researchers: high body weight (including obese patients, defined as BMI> 30 kg/m2), hypo-albuminaemia, clearance pathways, impact of extracorporeal clearance system (ECMO, CVVH).
exposure | 17 days
  To determine whether adequate exposure is attained in ICU patients
number of adverse events | 17 days
  To determine the safety of micafungin in this patient population

CONTACTS AND LOCATIONS:
Overall Officials: R Bruggemann, Principal Investigator — Radboud University Medical Center
Locations (4):
- Netherlands (4):
  - Rijstate Hospital, Arnhem
  - Gelderse Vallei Hospital, Ede
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Radboud University Nijmegen Medical Centre, Nijmegen

REFERENCES:
- [Result] Lempers VJ, Schouten JA, Hunfeld NG, Colbers A, van Leeuwen HJ, Burger DM, Verweij PE, Pickkers P, Bruggemann RJ. Altered Micafungin Pharmacokinetics in Intensive Care Unit Patients. Antimicrob Agents Chemother. 2015 Aug;59(8):4403-9. doi: 10.1128/AAC.00623-15. Epub 2015 May 11. PMID 25963988